CLINICAL TRIAL: NCT01746537
Title: Automated Analysis of Anterior Chamber Inflammation by Optical Coherence Tomography
Brief Title: Analysis of Anterior Chamber Inflammation by Optical Coherence Tomography
Acronym: ATAC
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Sunil Srivastava, Medical Doctor, The Cleveland Clinic
Other Study IDs: 12-612
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, observational, case series investigating the feasibility of utilizing OCT scans of the anterior chamber of eyes with uveitis.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Cole Eye Institute with uveitis.

Exclusion Criteria:

* Inability to provide informed consent, including non-English speaking and cognitively/mentally impaired.
* Severe corneal opacities preventing imaging of anterior chamber

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inactive and active uveitis.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-06; Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Use the OCT to objectively image and grade the degree of anterior chamber inflammation in eyes with inactive and active uveitis. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K Srivastva, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No